CLINICAL TRIAL: NCT00768157
Title: Efficacy of Antiviral Therapy With Lamivudine or Entecavir After Radical Resection for Hepatitis B Virus-Related Hepatocellular Carcinoma
Brief Title: Efficacy of Antiviral Therapy After Radical Resection for Hepatitis B Virus-Related Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Cancer Center of Sun Yat-sen University, Cancer Center of Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC-HCC004
Record Dates: First submitted 2008-10-06; First posted 2008-10-07 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2009-02

CONDITIONS: Hepatocellular Carcinoma; Hepatitis B Virus; Recurrence
Keywords: hepatocellular carcinoma; hepatitis B virus; surgery; anti-virus; recurrence
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hepatitis B; Recurrence | interventions — Lamivudine; entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- antiviral group (Experimental): Drug: antiviral treatment(lamivudine or entecavir) after the Procedure/Surgery (radical resection of HBV-related HCC)
  Interventions: Drug: antiviral treatment (lamivudine or entecavir); Procedure: radical resection of HBV-related HCC
- control group (Active Comparator): Procedure/Surgery (radical resection of HBV-related HCC) without Drug of antiviral treatment - close observation without antiviral treatment
  Interventions: Procedure: radical resection of HBV-related HCC

INTERVENTIONS:
Drug: antiviral treatment (lamivudine or entecavir) — antiviral treatment (lamivudine 100mg per day or entecavir 0.5mg per day)
  Arms: antiviral group
Procedure: radical resection of HBV-related HCC — Procedure/Surgery - radical resection of HBV-related HCC

SUMMARY:
Most hepatocellular carcinomas are associated with hepatitis B virus, it is hypothesized that anti-viral treatment may be helpful in treating HBV-related hepatocellular carcinoma.

DETAILED DESCRIPTION:
As we know, recurrence and metastasis could happen in hepatocellular carcinoma even after radical resection.One reason is that virus hepatitis B could be one factor contributing to the carcinogenesis of hepatocellular carcinoma.To investigated whether anti-viral therapy could improve the efficacy of radical resection of hepatitis B virus (HBV)-related hepatocellular carcinoma(HCC),we planed to conduct this clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. patients who did not receive antiviral therapy prior to the resection of hepatocellular carcinoma
2. patients who underwent radical resection of HCC, and 1 month after surgery,dynamic computed tomography showed on lesion in the liver and no signs of extrahepatic metastasis.
3. hepatitis B surface antigen should be positive before surgery HBV-DNA level between 100000 copies/ml and 10000000copies/ml anti-HCV negative

Exclusion Criteria:

1. previous history of antiviral therapy
2. a baseline serum alanine aminotransferase level 2.5 times the ULN or higher
3. positive for anti-HCV or anti-HIV
4. Child-Pugh classification B or C after surgery
5. preexisting evidence of hepatic decompensation, including encephalopathy,ascites,a bilirubin level more than 2 times the ULN, or a prolonged prothrombin time of more than 3 seconds
6. signs showing recurrence or metastasis oen month after surgery
7. underlying cardiac or renal diseases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2007-04; Primary Completion 2009-08 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
Overall survivals | 2,3,5years

SECONDARY OUTCOMES:
Recurrence rate | 2,3,5years

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Qing LI, Ph.D, Principal Investigator — Sun Yat-sen University; Min-Shan CHEN, Ph.D, Study Director — Sun Yat-sen University; Xiao-Jun LIN, Ph.D, Study Director — Sun Yat-sen University; Xiang-Ming LAO, Ph.D, Study Chair — Sun Yat-sen University
Locations (1):
- Xiang-Ming Lao, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Jang JW, Choi JY, Bae SH, Yoon SK, Chang UI, Kim CW, Cho SH, Han JY, Lee YS. A randomized controlled study of preemptive lamivudine in patients receiving transarterial chemo-lipiodolization. Hepatology. 2006 Feb;43(2):233-40. doi: 10.1002/hep.21024. PMID 16440357
- [Background] Jang JW, Choi JY, Bae SH, Yoon SK, Woo HY, Chang UI, Kim CW, Nam SW, Cho SH, Yang JM, Lee CD. The impact of hepatitis B viral load on recurrence after complete necrosis in patients with hepatocellular carcinoma who receive transarterial chemolipiodolization: implications for viral suppression to reduce the risk of cancer recurrence. Cancer. 2007 Oct 15;110(8):1760-7. doi: 10.1002/cncr.22984. PMID 17724708
- [Background] Jang JW, Choi JY, Bae SH, Kim CW, Yoon SK, Cho SH, Yang JM, Ahn BM, Lee CD, Lee YS, Chung KW, Sun HS. Transarterial chemo-lipiodolization can reactivate hepatitis B virus replication in patients with hepatocellular carcinoma. J Hepatol. 2004 Sep;41(3):427-35. doi: 10.1016/j.jhep.2004.05.014. PMID 15336446
- [Background] Poon RT. Significance of viral status on prognosis after resection of hepatitis B virus related hepatocellular carcinoma. J Hepatol. 2007 Nov;47(5):630-1. doi: 10.1016/j.jhep.2007.08.007. Epub 2007 Sep 5. No abstract available. PMID 17881079
- [Background] Sun HC, Zhang W, Qin LX, Zhang BH, Ye QH, Wang L, Ren N, Zhuang PY, Zhu XD, Fan J, Tang ZY. Positive serum hepatitis B e antigen is associated with higher risk of early recurrence and poorer survival in patients after curative resection of hepatitis B-related hepatocellular carcinoma. J Hepatol. 2007 Nov;47(5):684-90. doi: 10.1016/j.jhep.2007.06.019. Epub 2007 Aug 13. PMID 17854945
- [Background] Kubo S, Hirohashi K, Yamazaki O, Matsuyama M, Tanaka H, Horii K, Shuto T, Yamamoto T, Kawai S, Wakasa K, Nishiguchi S, Kinoshita H. Effect of the presence of hepatitis B e antigen on prognosis after liver resection for hepatocellular carcinoma in patients with chronic hepatitis B. World J Surg. 2002 May;26(5):555-60. doi: 10.1007/s00268-001-0267-1. Epub 2002 Feb 19. PMID 12098045
- [Background] Kubo S, Nishiguchi S, Hamba H, Hirohashi K, Tanaka H, Shuto T, Kinoshita H, Kuroki T. Reactivation of viral replication after liver resection in patients infected with hepatitis B virus. Ann Surg. 2001 Jan;233(1):139-45. doi: 10.1097/00000658-200101000-00020. PMID 11141236